CLINICAL TRIAL: NCT06464042
Title: Influence of Air Quality on the Development and Progression of Premature Coronary Artery Disease
Acronym: AIRHEART
Status: Recruiting | Type: Observational
Sponsor: pablo Juan-Salvadores (Other)
Collaborators: Fundacin Biomedica Galicia Sur (Other); Conselleria de Saúde Pública de Galicia (Unknown); Conselleria de Medio Ambiente, Territorio e Vivenda de Galicia (Unknown)
Responsible Party: Sponsor-Investigator, pablo Juan-Salvadores, Principal Investigator, Fundacin Biomedica Galicia Sur
Organization: Fundacin Biomedica Galicia Sur (Other)
Other Study IDs: AirHeart Study; SEC/FEC-INV-CLI 23/23 (Other Grant/Funding Number: Spanish Society of Cardiology); CI23-06 (Other Grant/Funding Number: Instituto de Investigación Sanitaria Galicia Sur)
Record Dates: First submitted 2024-06-03; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease Premature; Angina, Stable; Acute Coronary Syndrome; MINOCA; Myocardial Infarction
Keywords: Air pollution; young; Coronary Artery Disease Premature
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome; MINOCA; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature Coronary Artery Disease: Patients between 18 and 40 years old diagnosed with coronary artery disease, including: ST-elevation myocardial infarction (STEMI), non-ST-elevation acute coronary syndrome (NSTE-ACS), unstable angina, stable angina, MINOCA or silent angina
- Non Coronary Artery Disease: Patient without coronary artery disease
  For each case, 3 controls matched by age (±1 year), sex, postal code, and/or primary care center will be included. To avoid the selection of controls that could be associated with an overestimation of exposure to cardiovascular risk factors, the controls will be recruited from the preoperative unit and selected from subjects who have undergone minor clinical procedures (vasectomy, hernia repair, phimosis, prominent ear correction, tubal ligation, euthyroid thyroid nodule, plastic surgery, lipomas, vocal cord cysts, among others), or from the trauma service, selecting those attending for fractures or sprains. This approach ensures a complete medical history along with analytical values in their electronic medical records

SUMMARY:
The new global guidelines from the World Health Organization on air quality provide evidence of the damage that air pollution inflicts on human health at even lower concentrations than previously thought. Different studies have shown an increase in the incidence of coronary artery disease (CAD) in young people in recent decades. The main objective of this project is to study the impact of environmental pollutants on the premature manifestation of CAD from different epidemiological approaches and their impact on the evolution of these patients with a gender perspective. It is a retrospective analytical case-control study nested in a cohort of patients ≤40 years old with a clinical history of CAD including: ST-segment elevation myocardial infarction, non-ST-segment elevation acute coronary syndrome, unstable angina, stable angina or silent angina according to the international classification of diseases.

ELIGIBILITY:
CASES:

Inclusion Criteria:

* Women and men between 18 and 40 years old with a diagnosis of coronary artery disease coded in their medical records in Galicia

Exclusion Criteria:

* Not having a postal code and primary care center assigned in their medical records in Galicia

CONTROL

Inclusion Criteria:

* Women and men between 18 and 40 years old with no diagnosis or history of CAD or other coronary disease coded in their medical records

Exclusion Criteria:

* Present with non-ischemic coronary diseas.
* Have a serious condition that affects or decreases life expectancy.
* Do not have a postal code or primary care center assigned in their medical records in Galicia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study focuses on patients aged ≤40 years with a diagnosis of coronary artery disease (CAD) recorded in the clinical history of Galicia (IANUS), including: ST-elevation myocardial infarction (STEMI), non-ST-elevation acute coronary syndrome (NSTACS), unstable angina, stable angina, or silent angina according to the International Classification of Diseases (ICD-10). Given the limited number of cases, to increase the statistical power of the project, three patients without a diagnosis of CAD (controls) will be used for each patient with CAD confirmed by coronary angiography (case), matched by postal code and primary care center.
Sampling Method: Non-Probability Sample
Enrollment: 4272 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the differences in exposure to environmental pollutants in patients ≤40 years old with and without coronary artery disease | 15 years
  The study will measure the levels of environmental pollutants (such as PM2.5, PM10, nitrogen dioxide (NO2), carbon monoxide (CO), and ozone (O3), among others) in patients ≤40 years old with a clinical diagnosis of coronary artery disease and in patients without a diagnosis of coronary artery disease, in order to compare the differences.
To evaluate the impact of environmental pollutants on the incidence of the combined variable of major adverse cardiovascular events (MACE) up to 1, 5, and 10 years from the index cas | 15 years
  To evaluate the impact of environmental pollutants on the incidence of the combined variable of major adverse cardiovascular events (MACE) up to 1, 5, and 10 years from the index cas
To describe the prevalence of CAD in patients ≤40 years old in Galicia | 15 years
  To describe the prevalence of CAD in patients ≤40 years old in Galicia

SECONDARY OUTCOMES:
To evaluate the influence of PM2.5 and PM10 particles on the early manifestation of CAD. | 15 years
  The study will measure the levels of PM2.5, PM10 in patients ≤40 years old with a clinical diagnosis of coronary artery disease and in patients without a diagnosis of coronary artery disease, in order to compare the differences.
To describe the prevalence of ozone (O3), nitrogen dioxide (NO2), sulfur dioxide (SO2), benzene (C6H6), carbon monoxide (CO), and heavy metals such as arsenic, cadmium, nickel, and lead in the premature manifestation of CAD. | 15 years
  To describe the prevalence of ozone (O3), nitrogen dioxide (NO2), sulfur dioxide (SO2), benzene (C6H6), carbon monoxide (CO), and heavy metals such as arsenic, cadmium, nickel, and lead in the premature manifestation of CAD.
To determine the correlation of noise pollution with premature CAD by age and sex. | 15 years
  To determine the correlation of noise pollution with premature CAD by age and sex.
To identify the impact of temperatures on early CAD by age and sex. | 15 years
  The study will determine the impact of extreme temperatures, both heat and cold, on the premature presentation of coronary artery disease, by comparing this exposure between patients with and without the disease and sex.
To determine the correlation of environmental pollutants in patients with myocardial infarction with non-obstructive coronary arteries (MINOCA). | 15 years
  To determine the correlation of environmental pollutants in patients with myocardial infarction with non-obstructive coronary arteries (MINOCA).
To compare the effect of environmental pollutants and their relationship with CAD between men and women. | 15 years
  The influence of different environmental pollutants on the premature presentation of coronary artery disease will be analyzed, taking into account the differences between women and men.
To evaluate the incidence of serious adverse events | 15 years
  To evaluate the incidence of recurrent myocardial infarction, revascularizations (unplanned after admission), stroke, death, major bleeding (BARC scale 2 or higher), hospital admission for stable angina, unstable angina, acute coronary syndrome with or without ST elevation, congestive heart failure (CHF), or heart transplant during 1, 5, and 10 years. By age and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Juan-Salvadores, Pharma, PhD, Principal Investigator — Instituto de Investigación Sanitaria Galicia Sur (IIS Galicia Sur)
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juan-Salvadores P, Veiga C, Jimenez Diaz VA, Guitian Gonzalez A, Iglesia Carreno C, Martinez Reglero C, Baz Alonso JA, Caamano Isorna F, Romo AI. Using Machine Learning Techniques to Predict MACE in Very Young Acute Coronary Syndrome Patients. Diagnostics (Basel). 2022 Feb 6;12(2):422. doi: 10.3390/diagnostics12020422. PMID 35204511
- [Background] Juan-Salvadores P, Jimenez Diaz VA, Iglesia Carreno C, Guitian Gonzalez A, Veiga C, Martinez Reglero C, Baz Alonso JA, Caamano Isorna F, Iniguez Romo A. Coronary Artery Disease in Very Young Patients: Analysis of Risk Factors and Long-Term Follow-Up. J Cardiovasc Dev Dis. 2022 Mar 11;9(3):82. doi: 10.3390/jcdd9030082. PMID 35323630
- [Background] Juan-Salvadores P, Jimenez Diaz VA, Rodriguez Gonzalez de Araujo A, Iglesia Carreno C, Guitian Gonzalez A, Veiga Garcia C, Baz Alonso JA, Caamano Isorna F, Iniguez Romo A. Clinical Features and Long-Term Outcomes in Very Young Patients with Myocardial Infarction with Non-Obstructive Coronary Arteries. J Interv Cardiol. 2022 Jul 30;2022:9584527. doi: 10.1155/2022/9584527. eCollection 2022. PMID 35990214
- [Result] Chen R, Yin P, Meng X, Liu C, Wang L, Xu X, Ross JA, Tse LA, Zhao Z, Kan H, Zhou M. Fine Particulate Air Pollution and Daily Mortality. A Nationwide Analysis in 272 Chinese Cities. Am J Respir Crit Care Med. 2017 Jul 1;196(1):73-81. doi: 10.1164/rccm.201609-1862OC. PMID 28248546
- [Result] Orellano P, Reynoso J, Quaranta N, Bardach A, Ciapponi A. Short-term exposure to particulate matter (PM10 and PM2.5), nitrogen dioxide (NO2), and ozone (O3) and all-cause and cause-specific mortality: Systematic review and meta-analysis. Environ Int. 2020 Sep;142:105876. doi: 10.1016/j.envint.2020.105876. Epub 2020 Jun 23. PMID 32590284
- [Result] Kirwa K, Szpiro AA, Sheppard L, Sampson PD, Wang M, Keller JP, Young MT, Kim SY, Larson TV, Kaufman JD. Fine-Scale Air Pollution Models for Epidemiologic Research: Insights From Approaches Developed in the Multi-ethnic Study of Atherosclerosis and Air Pollution (MESA Air). Curr Environ Health Rep. 2021 Jun;8(2):113-126. doi: 10.1007/s40572-021-00310-y. PMID 34086258
- [Result] Chen SY, Hwang JS, Chan CC, Wu CF, Wu C, Su TC. Urban Air Pollution and Subclinical Atherosclerosis in Adolescents and Young Adults. J Adolesc Health. 2022 Aug;71(2):233-238. doi: 10.1016/j.jadohealth.2022.03.004. Epub 2022 May 7. PMID 35537887
- See also: Video — https://youtu.be/eXlTfhdBByA